CLINICAL TRIAL: NCT01689597
Title: Efficacy of Two Doses of Epidural Morphine for Analgesia After Traumatic Vaginal Delivery: a Randomized, Double Blinded, Placebo-controlled Pilot Study
Brief Title: Epidural Morphine for Analgesia After Traumatic Vaginal Delivery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn - no participants enrolled
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18501
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2012-09

CONDITIONS: Traumatic Vaginal Delivery
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose epidural morphine (Active Comparator): One dose of 1.25 mg epidural morphine
  Interventions: Drug: Morphine
- High dose epidural morphine (Active Comparator): One dose of 2.5 mg epidural morphine
  Interventions: Drug: Morphine
- Saline (Placebo Comparator): One dose of 10 ml saline administered through an epidural catheter
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine — Comparison of different dosages of drug
  Arms: High dose epidural morphine; Low dose epidural morphine
Drug: Placebo
  Arms: Saline

SUMMARY:
This pilot study intends to establish the efficacy of 2 different doses of epidural morphine for pain management after perineal trauma when using multimodal analgesia as well as the feasibility of conducting a larger randomized clinical trial. Women with traumatic vaginal delivery will be randomized into 3 groups with 10 patients each and receive 2.5 mg epidural morphine, 1.25 mg epidural morphine, or epidural saline. The primary outcome is total opioid consumption for breakthrough pain in the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 years or older
* The patient is ASA 1-3
* Gestation 37-42 weeks
* The patient had a vaginal delivery
* The patient received epidural analgesia for labor and delivery

Exclusion Criteria:

* The patient has refused to participate
* The patient cannot give informed consent
* The investigator has significant concerns for maternal or neonatal welfare
* The patient has a history of allergy to opioids
* The patient has a history of chronic opioid consumption
* The patient has a history of narcotic abuse
* The patient has an allergy to local anesthetics
* The patient has a contraindication to taking NSAIDs or acetaminophen
* The patient received combined spinal-epidural analgesia
* The patient has a history of chronic pain

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09 (Estimated); Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Total breakthrough opioid consumption | First 24 hours after delivery

SECONDARY OUTCOMES:
Pain scores at rest | At 6, 12, 24, and 36 h after delivery
Pain scores with movement | At 6, 12, 24, and 36 h after delivery
Severity of nausea/vomiting | At 6, 12, 24, and 36 h after delivery
Severity of pruritis | At 6, 12, 24, and 36 h after delivery
Severity of sedation | At 6, 12, 24, and 36 h after delivery
Time to first request for additional analgesia | First 36 h after delivery
Patient satisfaction with pain control | At 24 and 36 h after delivery
Quality of Recovery | At 24 and 36 h after delivery
Antiemetic consumption | First 36 h after delivery
Antipruritic medication consumption | First 36 h after delivery
Total opioid consumption | First 36 h after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sudha I Singh, MD FRCPC, Principal Investigator — The University of Western Ontario